CLINICAL TRIAL: NCT02356783
Title: Implementation of Wireless Pedometer for Monitoring Step Count Before and After Lumbar Epidural Steroid Injection for Radicular Pain.
Brief Title: Implementation of Pedometer for Monitoring Step Count Pre and Post Lumbar ESI for Radicular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: #2014-135
Record Dates: First submitted 2015-01-13; First posted 2015-02-05 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interlaminar (Other): Approach for lumbar epidural steroid injection for this arm will be interlaminar.
  We will be implementing a wireless pedometer to each of the 15 patients in this group to measure our primary and secondary outcomes.
  Interventions: Device: Pedometer
- Transforaminal (Other): Approach for lumbar epidural steroid injection for this arm will be transforaminal.
  We will be implementing a wireless pedometer to each of the 15 patients in this group to measure our primary and secondary outcomes.
  Interventions: Device: Pedometer

INTERVENTIONS:
Device: Pedometer — Wireless pedometer

SUMMARY:
Our aim is to assess usability and compliance of a wireless pedometer for monitoring step count after a lumbar epidural steroid injection for the treatment of radicular pain in low back pain patients. Our main hypothesis is to demonstrate pedometer measured step count can be used to measure efficacy of pain interventions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Patients receiving lumbar epidural steroid injections as pain management to be scheduled at least one week away (-2 days/1 month).
* Patients who are able to understand how the Fitbit instrument works and are willing to consent to the study.
* Patient who used web-based communication frequently, e.g. Email.
* Patients who can speak, understand, and write in English.
* Prior MRI or an appointment to obtain an MRI prior to the procedure.

Exclusion Criteria:

* Workers' compensation cases.
* Patient does not have a computer at home.
* Non-ambulatory patients.
* Patients who have received a lumbar epidural steroid injection in the past 6 months.
* Nursing or pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Griffin, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital For Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Cohen SP, Bicket MC, Jamison D, Wilkinson I, Rathmell JP. Epidural steroids: a comprehensive, evidence-based review. Reg Anesth Pain Med. 2013 May-Jun;38(3):175-200. doi: 10.1097/AAP.0b013e31828ea086. PMID 23598728
- [Background] MacVicar J, King W, Landers MH, Bogduk N. The effectiveness of lumbar transforaminal injection of steroids: a comprehensive review with systematic analysis of the published data. Pain Med. 2013 Jan;14(1):14-28. doi: 10.1111/j.1526-4637.2012.01508.x. Epub 2012 Oct 30. PMID 23110347

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-three patients were enrolled in study and received FitBit prior to their steroid injection appointment. Only 33 patients returned to have the steroid injection (16 interlaminar, 17 transforaminal). Three transforaminal and 1 interlaminar patient stopped using/syncing the FitBit, so data were not available to analyze.
Groups:
- Interlaminar: Approach for lumbar epidural steroid injection for this arm will be interlaminar.
  We will be implementing a wireless pedometer to each of the 15 patients in this group to measure our primary and secondary outcomes.
  Pedometer: Wireless pedometer
- Transforaminal: Approach for lumbar epidural steroid injection for this arm will be transforaminal.
  We will be implementing a wireless pedometer to each of the 15 patients in this group to measure our primary and secondary outcomes.
  Pedometer: Wireless pedometer
Period: Overall Study
Arm/Group | Interlaminar | Transforaminal
Started | 16 | 17
Completed | 15 | 14
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interlaminar | Transforaminal | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (16.2) | 51.5 (12.9) | 53.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 5 | 7 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Available Step Count Data at Baseline.
Description: Percentage of patients with available step count data 7 days pre-procedure. Step count will be obtained daily for 7 days using a wireless pedometer.
Time Frame: A week pre-procedure.
Measure: Number; unit: percentage of patients with step data
Arm/Group | Interlaminar | Transforaminal
Number analyzed (Participants) | 15 | 14
percentage of patients with step data | 93.3 | 71.4

2. Primary Outcome: Percentage of Patients With Available Step Count Data Post-procedure.
Description: Percentage of patients with available step count data 60 days post-procedure. Step count will be obtained using a wireless pedometer daily for a period of 60 days post-procedure.
Time Frame: Duration of 60 days after procedure.
Measure: Number; unit: percentage of patients with step data
Arm/Group | Interlaminar | Transforaminal
Number analyzed (Participants) | 15 | 14
percentage of patients with step data | 73.3 | 57.1

ADVERSE EVENTS:
Arm/Group | Interlaminar | Transforaminal
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes